CLINICAL TRIAL: NCT06893991
Title: The Effect of Symbiotic Beverage Consumption on Lipid Profile and Nutritional Status in Overweight and Hypercholesterolemia Adults Aged Above 18 Years
Brief Title: The Effect of Symbiotic Beverage Consumption on Lipid Profile
Acronym: SYMBIONIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Politeknik Kesehatan Kemenkes Padang (Other)
Responsible Party: Principal Investigator, Gusnedi, Associate Professor, Dr, Politeknik Kesehatan Kemenkes Padang
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PoliteknikKKP
Record Dates: First submitted 2025-03-05; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Lipid Profile; Fasting Blood Sugar Above Normal; Body Mass Index
Keywords: Symbiotic Beverages; Lipid Profile; Body Mass Index
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This trial is a controlled clinical studies conducted to evaluate the effectiveness of the symbiotic drink for improving lipid profiles, blood sugar and nutritional status in participants with hypercholesterolemia or overweight under study and to determine the common short-term side effects and risks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Consuming 100 ml Symbiotic beverages every day for 6 weeks plus dietary advice to overcome dyslipidemia
  Interventions: Dietary Supplement: SYMBIONIC; Behavioral: Dietary advice
- Comparison group (Active Comparator): Receiving standard dietary advice to overcome dyslipidemia, but without drinking symbiotic beverage
  Interventions: Behavioral: Dietary advice

INTERVENTIONS:
Dietary Supplement: SYMBIONIC — Provision of 100 ml symbiotic beverages "daygurt" per day for 6 weeks, plus standard dietary advice for dyslipidemia
  Arms: Intervention Group
Behavioral: Dietary advice — Participants get standard dietary advice for dyslipidemia

SUMMARY:
The goal of this clinical trial is to evaluate whether the synbiotic beverage "Daygurt" can improve lipid profiles, blood sugar levels, blood pressure, and body weight in individuals diagnosed with dyslipidemia. The main questions it aims to answer are:

Does "Daygurt" significantly reduce total cholesterol and LDL levels compared to nutrition counseling alone? Does "Daygurt" increase HDL levels and reduce triglycerides more effectively than nutrition counseling? Does "Daygurt" lead to greater improvements in fasting blood sugar, blood pressure, and body weight compared to nutrition counseling?

The intervention group (receiving "Daygurt" plus nutrition counseling) will be compared to the comparison group (receiving nutrition counseling without "Daygurt") to see if "Daygurt" provides additional benefits beyond standard dietary advice.

Participants will be divided into 2 groups:

Intervention group: Consume "Daygurt" daily for 8 weeks. Comparison group: Receive nutrition counseling sessions focused on managing dyslipidemia but will not consume "Daygurt."

Both groups will undergo health parameter measurements before and after the intervention, including:

Total cholesterol, LDL, HDL, and triglyceride levels. Fasting blood sugar. Blood pressure. Body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* Cholesterol total above 200 mg/dl, or LDL Cholesterol above 100, or BMI above 25 kg/m2
* Agree to study protocols

Exclusion Criteria:

* Has Allergic to dairy product
* Having any drug lowering cholesterol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 6 weeks (before and after intervention)
  Fasting Total blood cholesterol, LDL cholesterol, HDL cholesterol and triglyceride level measured before and after intervention phase

CONTACTS AND LOCATIONS:
Locations (1):
- Health Ministry Polytechnic of Padang, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided